CLINICAL TRIAL: NCT06592222
Title: Comparative Effectiveness of Elranatamab in Clinical Study C1071003 Versus Physician's Choice of Treatment (PCT) in Real-World (RW) External Control Arms in Patients With Triple-Class Refractory (TCR) Multiple Myeloma (MM)
Brief Title: A Study to Learn About the Effectiveness of the Medicine Called Elranatamab in People With Relapsed Refractory Multiple Myeloma as Compared With Standard of Care Therapies
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1071043
Record Dates: First submitted 2024-08-08; First posted 2024-09-19 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elranatamab: Patients treated with elranatamab from the MagnetisMM-3 trial
  Interventions: Drug: Elranatamab
- Standard of care: Patients treated with standard-of-care therapies from real-world data sources
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Elranatamab — BCMA-CD3 bispecific antibody
  Groups: Elranatamab
Drug: Standard of care — Standard of care
  Groups: Standard of care

SUMMARY:
This study is to understand how well elranatamab (PF-06863135) may be used for relapsed refractory multiple myeloma (RRMM). Sometimes MM might improve at first, but then gets resistant to the treatment and starts growing again (known as relapsed refractory). This study medicine will be compared with standard-of-care (SOC) therapies used in real-world clinical practice. For people receiving elranatamab, the investigators will use data from the phase 2 clinical trial (MagnetisMM-3). The investigators will also use data from a real-world data source, representing the SOC in clinical practice. This study does not seek any participants for enrollment. The investigators will compare the experiences of people receiving elranatamab to people receiving SOC therapies. This way, it will help the investigators to know how well elranatamab can be used for RRMM treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older at index date
* Diagnosis of MM
* Measurable disease according to IMWG criteria
* ECOG performance status ≤2
* Refractory to at least 1 proteasome inhibitor, 1 immunomodulatory drug, and 1 anti-CD38 treatment (ie, triple-class refractory [TCR])
* At least 1 treatment following their TCR eligibility

Exclusion Criteria:

* Acute plasma cell leukemia
* Amyloidosis
* Smoldering MM
* Stem cell transplant within 12 weeks of index or active graft versus host disease (GVHD)
* Active malignancy within 3 years before index, except for basal cell or squamous cell skin cancer or carcinoma in situ
* Administration with an investigational drug within 30 days prior to index

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with elranatamab will come from the MagnetisMM-3 trial. Patients treated with the standard-of-care therapies will come from real-world data sources.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From the index therapy start until progression or death due to any cause, whichever occurs first, assessed up to 6 years

SECONDARY OUTCOMES:
Overall surival | From the index therapy start until death due to any cause assessed up to 6 years
Duration of response | From the first documentation of objective response until progression or death due to any cause, whichever occurs first, assessed up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071043